CLINICAL TRIAL: NCT01691911
Title: Preconditioning Shields Against Vascular Events in Surgery. A Multi-Centre Trial of Preconditioning Against Adverse Events in Major Vascular Surgery
Brief Title: Preconditioning Shields Against Vascular Events in Surgery
Acronym: SAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Professor Stewart Walsh, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAVES-123
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Abdominal Aortic Aneurysm; Carotid Atherosclerosis; Critical Lower Limb Ischaemia
Keywords: Vascular disease; Open aortic aneurysm repair; Endovascular aneurysm repair; Carotid endartrectomy; Lower limb surgical revascularisation; Major lower limb amputation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Carotid Artery Diseases; Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote preconditioning (Experimental): Preconditioning will be performed in the same manner as several previous trials. Immediately after induction of anaesthesia, a standard, CE-approved blood pressure cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 4 ischaemia-reperfusion cycles. In all other respects, the procedure and peri-operative care will follow the routine practices of the surgeons and anaesthetists involved.
  Interventions: Procedure: Remote preconditioning
- Remote preconditioning control (No Intervention): Patients randomised to this group will receive routine pre-operative, peri-operative and post operative care.

INTERVENTIONS:
Procedure: Remote preconditioning — Immediately after induction of anaesthesia, a standard, CE-approved tourniquet cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 4 ischaemia-reperfusion cycles. In all other respects, the procedure and peri-operative care will follow the routine practices of the surgeons and anaesthetists involved.
  Arms: Remote preconditioning

SUMMARY:
Major vascular surgery involves operations to repair swollen blood vessels, clear debris from blocked arteries or bypass blocked blood vessels. Patients with these problems are a high-risk surgical group as they have generalized blood vessel disease. These puts them at risk of major complications around the time of surgery such as heart attacks , strokes and death. The mortality following repair of a swollen main artery in the abdomen is about 1 in 20. This contrasts poorly with the 1 per 100 risk of death following a heart bypass. Simple and cost-effective methods are needed to reduce the risks of major vascular surgery. Remote ischaemic preconditioning (RIPC) may be such a technique. To induce RIPC, the blood supply to muscle in the patient's arm is interrupted for about 5 minutes. It is then restored for a further five minutes. This cycle is repeated three more times. The blood supply is interrupted simply by inflating a blood pressure cuff to maximum pressure. This repeated brief interruption of the muscular blood supply sends signals to critical organs such as the brain and heart, which are rendered temporarily resistant to damage from reduced blood supply. Several small randomized clinical trials in patients undergoing different types of major vascular surgery have demonstrated a potential benefit. This large, multi-centre trial aims to determine whether RIPC can reduce complications in routine practice.

DETAILED DESCRIPTION:
The demand for major vascular surgery is increasing [1]. Patients requiring procedures such as aortic aneurysm repair, carotid endarterectomy, lower limb surgical re-vascularisation and major lower limb amputation for end-stage vascular disease constitute a high-risk surgical cohort. Peri-operative complications such as myocardial infarction, cerebrovascular accident, renal failure and death are common [2,3]. Multiple potential mechanisms may result in these complications. For example, myocardial injury may result from systemic hypotension leading to reduced flow across a tight coronary artery stenosis or, alternatively, it may arise due to acute occlusion when an unstable plaque ruptures. Most strategies aimed at peri-operative risk reduction target a single potential mechanism. For example, beta-blockade may prevent myocardial injury due to overwork, but cannot prevent acute coronary occlusion. There is a requirement for a simple, effective intervention that protects tissues against injury via multiple different mechanisms. Remote ischemic preconditioning (RIPC) may be suitable.

Ischemic preconditioning is a phenomenon whereby a brief period of non-lethal ischemia in a tissue renders it resistant to the effects of a subsequent much longer ischaemic insult. It was first described in the canine heart [4]. Subsequent clinical trials showed that ischemic preconditioning reduced heart muscle damage following coronary artery bypass grafting [5] and liver dysfunction following hepatic resection [6]. Following cardiac surgery, it is associated with a reduction in critical care stay, arrhythmias and inotrope use [7]. However, ischemic preconditioning requires direct interference with the target tissues' blood supply, limiting its clinical utility. Further experimental work suggested that brief ischemia in one tissue, such as the kidneys, could confer protection on distant organs such as the heart [8]. A similar effect was observed after transient skeletal muscle ischemia [9-11]. This effect is referred to as 'preconditioning at a distance' or 'remote ischemic preconditioning' (RIPC).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* patient willing to give full informed consent for participation
* Patients undergoing elective carotid endarterectomy or
* Patients undergoing open abdominal aortic aneurysm repair or
* Patients undergoing endovascular abdominal aneurysm repair or
* Patients undergoing surgical lower limb revascularisation (suprainguinal or infrainguinal)

Exclusion Criteria:

* Patients less than 18 years of age
* Patients who are unable or unwilling to give full informed consent
* Pregnancy
* Significant upper limb peripheral arterial disease
* Patients on glibenclamide or nicorandil (these medications may interfere with remote ischaemic preconditioning)
* Patients with an estimated pre-operative glomerular filtration rate < 30mls/min/1.73m2
* Patients with a history of myocarditis, pericarditis or amyloidosis
* Patients undergoing Fenestrated or branched EVAR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Major Adverse Clinical Events | 30 day
  The primary endpoint for the trial will be Major Adverse Clinical Events. This is a composite endpoint comprising any of: cardiovascular death, myocardial infarction, new onset arrhythmia requiring treatment, cardiac arrest, congestive cardiac failure, cerebrovascular accident, renal failure requiring renal replacement therapy, mesenteric ischaemia requiring intervention or biopsy proven ischaemic colitis, urgent cardiac revascularisation. All participants will undergo a serum troponin levels and 12-lead electrocardiogram on the second post-operative day to screen for silent peri-operative myocardial infarction. Trial ECGs and troponin levels will be interpreted by a blinded trial cardiologist.

SECONDARY OUTCOMES:
Duration of post-operative hospital stay | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Duration of intensive care unit stay | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Unplanned critical care unit admission | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Acute kidney injury score in first three peri-operative days | 3 days
  The Acute Kidney Injury Score will be calculated over the first three peri-operative days. Creatinine will be measured daily as part of routine care. Urine volumes will be calculated from the fluid balance charts maintained as part of usual care.
Peri-operative myocardial injury | from operation to 72 hours postoperatively
  Peri-operative myocardial injury will be assessed by measurement of serum troponin levels. This will be achieved by comparing area under the curve (AUC) for serum troponin concentration over the first three post-operative days.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart R Walsh, MCh FRCS, Principal Investigator — Mid Western Regional Hospital and University of Limerick
Locations (1):
- MidWestern Regional Hospital, Limerick, Limerick, Ireland

REFERENCES:
- [Background] Anderson PL, Gelijns A, Moskowitz A, Arons R, Gupta L, Weinberg A, Faries PL, Nowygrod R, Kent KC. Understanding trends in inpatient surgical volume: vascular interventions, 1980-2000. J Vasc Surg. 2004 Jun;39(6):1200-8. doi: 10.1016/j.jvs.2004.02.039. PMID 15192558
- [Background] Chambers BR, Donnan GA. Carotid endarterectomy for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD001923. doi: 10.1002/14651858.CD001923.pub2. PMID 16235289
- [Background] Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG; EVAR trial participants. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet. 2004 Sep 4-10;364(9437):843-8. doi: 10.1016/S0140-6736(04)16979-1. PMID 15351191
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Jenkins DP, Pugsley WB, Alkhulaifi AM, Kemp M, Hooper J, Yellon DM. Ischaemic preconditioning reduces troponin T release in patients undergoing coronary artery bypass surgery. Heart. 1997 Apr;77(4):314-8. doi: 10.1136/hrt.77.4.314. PMID 9155608
- [Background] Clavien PA, Selzner M, Rudiger HA, Graf R, Kadry Z, Rousson V, Jochum W. A prospective randomized study in 100 consecutive patients undergoing major liver resection with versus without ischemic preconditioning. Ann Surg. 2003 Dec;238(6):843-50; discussion 851-2. doi: 10.1097/01.sla.0000098620.27623.7d. PMID 14631221
- [Background] Walsh SR, Tang TY, Kullar P, Jenkins DP, Dutka DP, Gaunt ME. Ischaemic preconditioning during cardiac surgery: systematic review and meta-analysis of perioperative outcomes in randomised clinical trials. Eur J Cardiothorac Surg. 2008 Nov;34(5):985-94. doi: 10.1016/j.ejcts.2008.07.062. Epub 2008 Sep 9. PMID 18783958
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Birnbaum Y, Hale SL, Kloner RA. Ischemic preconditioning at a distance: reduction of myocardial infarct size by partial reduction of blood supply combined with rapid stimulation of the gastrocnemius muscle in the rabbit. Circulation. 1997 Sep 2;96(5):1641-6. doi: 10.1161/01.cir.96.5.1641. PMID 9315559
- [Background] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Background] Oxman T, Arad M, Klein R, Avazov N, Rabinowitz B. Limb ischemia preconditions the heart against reperfusion tachyarrhythmia. Am J Physiol. 1997 Oct;273(4):H1707-12. doi: 10.1152/ajpheart.1997.273.4.H1707. PMID 9362234
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250